CLINICAL TRIAL: NCT02443987
Title: Time Interval Between TVT and First Void (TIBT) Study
Acronym: TIBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gloucestershire Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 15/013/GHT
Record Dates: First submitted 2015-04-27; First posted 2015-05-14 (Estimated); Results first posted 2025-10-29 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2017-08

CONDITIONS: Stress Urinary Incontinence
Keywords: Tension-Free Vaginal Tape
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Received intravenous fluids (Experimental): The patient will receive 500ml of 0.9% NaCl fluid intravenously during the operation.
  Interventions: Other: Intravenous fluid
- Control Arm (No Intervention): The patient will receive no intravenous fluid as per current routine protocol

INTERVENTIONS:
Other: Intravenous fluid — 500ml infusion of 0.9% Sodium Chloride intravenously.
  Arms: Received intravenous fluids

SUMMARY:
The primary aim of this study is to compare, in women undergoing tension-free vaginal tape (TVT) insertion under sedation and local anaesthetic infiltration, the time interval of first void following surgery between a group of patients who received intravenous fluids to those who did not.

DETAILED DESCRIPTION:
Urinary incontinence is a global condition and its prevalence increases with age. It impairs quality of life of patients and has a significant burden on the health care system. Stress urinary incontinence (SUI) is defined as involuntary leakage of urine when there is an increase in pressure on the bladder, i.e. during exercise, coughing or sneezing. It is the commonest form of urinary incontinence and affects around 50% of women with symptoms of incontinence.

The development of mid urethral tapes (e.g. the tension free vaginal tape [TVT]) in 1998 has greatly changed clinical practice. The introduction of TVTs has reduced the average length of hospital stay for patients undergoing surgical treatment of SUI by over 50%. As a result, the hospital bed occupancy for the treatment of SUI has decreased by a similar amount. Studies have shown it to have similar effectiveness to the main alternative surgical treatments in SUI.

In Gloucestershire Royal Hospital, we perform the procedure as a daycase with local anaesthetic infiltration under sedation. Routine cystoscopy is performed as a part of the procedure to exclude bladder trauma. The bladder is emptied at the end of procedure. Patients are then allowed to drink as normal and post void residuals are checked before discharge to rule out any problems emptying the bladder. It has been observed that the major limiting factor in early discharge of patients is the time to first void following surgery. As the patients are starved for surgery, they are often dehydrated and therefore require enough oral fluids to rehydrate and fill their bladder in order to void. If we can somehow reduce this waiting period, we can discharge patients sooner improving their experience with the surgery. We would like to examine whether filling up the bladder intra-operatively with intravenous fluid will reduce this time limiting step.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study

Exclusion Criteria:

* TVT performed under general or spinal anaesthetic
* Women under the age of 18 years
* Women unable to give informed consent
* TVT performed in addition to another procedure
* Women not suitable for a fluid challenge due to co-morbidities.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2015-08; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark James, MBChB MD, Principal Investigator — Gloucestershire Hospitals NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - Gloucestershire Royal Hospital, Gloucester
  - Stroud General Hospital, Stroud

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment from October 2015 to June 2016. Recruited from urogynaecology clinic on decision to add to TVT waiting list.
Pre-assignment Details: 3 Patient's operations were cancelled by the surgeon or the patient prior to randomisation.
Groups:
- Received intravenous fluids: The patient received 500ml of 0.9% sodium chloride fluid intravenously during the operation.
- Control Arm: The patient received no intravenous fluid as per current routine protocol
Period: Overall Study
Arm/Group | Received intravenous fluids | Control Arm
Started | 23 | 20
Completed | 22 | 18
Not Completed | 1 | 2
Not completed — Bladder injury | 1 | 1
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Received intravenous fluids | Control Arm | Total
Number analyzed (Participants) | 22 | 18 | 40
Age, Customized [Count of Participants; unit: Participants]
  18 years or above | 22 | 18 | 40
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 22 | 18 | 40
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Time Interval Between End of Surgery and First Void
Time Frame: The participants will be followed for the duration of hospital stay, which is expected to be an average of 6 hours (and no longer than 24 hours)
Measure: Mean (Full Range); unit: minutes
Arm/Group | Received intravenous fluids | Control Arm
Number analyzed (Participants) | 22 | 18
minutes | 183 [30 to 420] | 197 [90 to 290]
Statistical Analysis 1: Comparison: Received intravenous fluids vs Control Arm; Test type: Superiority; p = 0.40, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Volume of Urine Passed
Description: Volume of urine passed at first void
Time Frame: as for outcome 1
Measure: Mean (Full Range); unit: mL
Arm/Group | Received intravenous fluids | Control Arm
Number analyzed (Participants) | 22 | 18
mL | 269 [21 to 600] | 199 [62 to 600]
Statistical Analysis 1: Comparison: Received intravenous fluids vs Control Arm; Test type: Superiority; p = 0.18, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Residual Volume in Bladder
Description: Residual volume of urine left in the bladder after first void as measured by bladder scanning
Time Frame: as for outcome 1
Measure: Mean (Full Range); unit: mL
Arm/Group | Received intravenous fluids | Control Arm
Number analyzed (Participants) | 22 | 18
mL | 141 [0 to 652] | 42 [0 to 220]
Statistical Analysis 1: Comparison: Received intravenous fluids vs Control Arm; Test type: Superiority; p = 0.02, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Time to "Fit for Discharge"
Description: Time interval between end of surgery to when staff deem patient is fit for discharge.
Time Frame: as for outcome 1
Measure: Mean (Full Range); unit: minutes
Arm/Group | Received intravenous fluids | Control Arm
Number analyzed (Participants) | 22 | 18
minutes | 355 [135 to 1443] | 339 [175 to 945]
Statistical Analysis 1: Comparison: Received intravenous fluids vs Control Arm; Test type: Superiority; p = 0.51, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Number of Patient's Requiring In-out Catheterisation Due to Difficulty Voiding
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Received intravenous fluids | Control Arm
Number analyzed (Participants) | 22 | 18
Participants | 2 | 0

6. Secondary Outcome: Patient Satisfaction Using Patient Questionnaire
Description: Patients were asked to grade their experience using a series of questions. They were asked to answer each on a scale of 0 to 10 in terms of satisfaction, with 0 = not at all and 10 = extremely (numbers 1-9 were not classified). Therefore the higher the score the more positive the patient experience.
Time Frame: as for outcome 1
Population: 2 patients did not return a completed satisfaction questionnaire.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Received intravenous fluids | Control Arm
Number analyzed (Participants) | 21 | 17
units on a scale
  Satisfaction with explanation | 9.9 [9 to 10] | 9.9 [9 to 10]
  Anxiety before | 6.5 [1 to 10] | 5.6 [0 to 10]
  Satisfied with explanation of discomfort | 9.4 [7 to 10] | 9.7 [7 to 10]
  Rating of support from staff during the procedure | 9.9 [8 to 10] | 9.8 [8 to 10]
  Satisfaction with privacy and dignity | 10.0 [10 to 10] | 9.8 [7 to 10]
  Satisfaction with length of stay | 9.0 [4 to 10] | 9.8 [9 to 10]
  Satisfaction with length of time to first void | 8.3 [2 to 10] | 8.7 [4 to 10]
  Overall satisfaction with procedure | 9.7 [8 to 10] | 9.9 [9 to 10]

ADVERSE EVENTS:
Time Frame: Adverse event data collected over 1 month post surgery.
Arm/Group | Received intravenous fluids | Control Arm
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/20
Other Adverse Events (participants affected / at risk) | 1/23 | 1/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Received intravenous fluids (N=23) | Control Arm (N=20)
Bladder injury (Renal and urinary disorders) | 1 | 1 — Bladder injury at time of surgery - related to the surgery and not directly due to study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes